CLINICAL TRIAL: NCT06872801
Title: Comparison of the Effects of Home High-Flow Nasal Cannula Therapy and Noninvasive Ventilation in Patients With Stable Chronic Hypercapnic Respiratory Failure
Brief Title: Home High-Flow Nasal Cannula vs. Noninvasive Ventilation for Stable Chronic Respiratory Failure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wonju Severance Christian Hospital (Other)
Responsible Party: Principal Investigator, Sang-Ha Kim, Professor, Wonju Severance Christian Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: WonjuSCH-SHK001-V1.0
Record Dates: First submitted 2025-02-26; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-04

CONDITIONS: Stable Chronic Hypercapnic Respiratory Failure
Keywords: Chronic Hypercapnic Respiratory Failure; Noninvasive Ventilation; High-Flow Nasal Cannula; Randomized Controlled Trial; Crossover Design
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- HFNC-NIV (Experimental): Participants first use HFNC for six weeks, then switch to NIV for six weeks
  Interventions: Device: High-Flow Nasal Cannula; Device: Noninvasive Ventilation
- NIV-HFNC (Experimental): Participants first use NIV for six weeks, then switch to HFNC for six weeks
  Interventions: Device: High-Flow Nasal Cannula; Device: Noninvasive Ventilation

INTERVENTIONS:
Device: High-Flow Nasal Cannula — To compare the effects of NIV (Trilogy Evo®) and HFNC (myAirvo2®) in patients with chronic hypercapnic COPD.
Device: Noninvasive Ventilation — to compare the effects of NIV (Trilogy Evo®) and HFNC (myAirvo2®) in patients with chronic hypercapnic COPD

SUMMARY:
The goal of this clinical trial is to compare the effects of home high-flow nasal cannula (HFNC) therapy and noninvasive ventilation (NIV) in patients with stable chronic hypercapnic respiratory failure. The main questions it aims to answer are:

* Does HFNC or NIV reduce blood carbon dioxide levels more effectively?
* How well do patients tolerate and adhere to each therapy?
* Are there differences in oxygen saturation, respiratory rate, and quality of life between the two treatments?

Participants Will:

* Use either HFNC (myAirvo2®) or NIV (Trilogy Evo®) every night for at least 4 hours over a 6-week period.
* Visit the hospital for checkups and arterial blood gas tests at the end of each 6-week period.
* Switch to the alternate device after six weeks as part of the crossover study design.
* Have their device usage recorded and analyzed.

DETAILED DESCRIPTION:
[Objectives and Background] Noninvasive ventilation (NIV) is the standard treatment for respiratory failure caused by acute exacerbations of chronic obstructive pulmonary disease (COPD). Numerous recent studies have demonstrated its efficacy, showing improvements in arterial blood gas results, reduced intubation rates, shorter hospital stays, and lower mortality rates.

Some studies suggest that NIV may also be beneficial for patients with stable chronic hypercapnic COPD. Randomized controlled trials (RCTs) have confirmed that applying NIV in these patients reduces one-year mortality, acute exacerbations, and hospital admission rates, while improving hypercapnia, oxygen saturation, respiratory rate, dyspnea, six-minute walk test results, and quality of life. However, some patients have difficulty adapting to NIV, limiting their benefits from the therapy.

High-flow nasal cannula (HFNC) therapy has been developed to deliver heated and humidified air through slightly enlarged nasal prongs. HFNC effectively reduces dead space by rapidly clearing expiratory gas from the upper airway and ensures the delivery of high-flow gas without dilution with ambient air. Studies have shown that HFNC reduces intubation rates and mortality in patients with severe hypoxemic respiratory failure. Compared to NIV, HFNC is not inferior in terms of re-intubation rates. Moreover, HFNC has demonstrated rapid reductions in CO2 levels in hypercapnic patients. Preliminary studies have confirmed its effectiveness in long-term use for patients with stable chronic hypoxemic or hypercapnic respiratory failure, with the most effective flow rates ranging from 30-50 L/min.

This clinical trial aims to compare the effects of NIV and HFNC (myAirvo2®) in patients with chronic hypercapnic COPD. Participants will use each device for six weeks in a crossover design, and the primary outcome will be a comparison of arterial CO2 reduction.

[Inclusion Criteria, Exclusion Criteria, Target Sample Size, and Rationale]

1. Inclusion Criteria:

   * Adults aged 40 years or older
   * Diagnosed with COPD
   * Resting arterial blood gas analysis showing pCO2 > 45 mmHg
   * Ability to read and write Korean
   * Voluntarily provided written informed consent For elderly patients (≥80 years), if cognitive function or judgment is impaired, informed consent may also be obtained from a legal representative. During the study period, participants will receive device training and explanations in a quiet setting to ensure understanding.
2. Exclusion Criteria:

   * Refusal to consent
   * Difficulty using NIV or HFNC
   * Cognitive impairment preventing understanding of the study
   * Acute exacerbation of hypoxemia or hypercapnia within the past four weeks
3. Target Sample Size: 38 Participants
4. Rationale for Sample Size: A previous study confirmed a significant reduction in arterial CO2 levels of 4 mmHg with HFNC compared to standard treatment in stable hypercapnic COPD patients. This study is designed as a non-inferiority crossover trial, with a non-inferiority margin of -4 mmHg, a standard deviation of 6.0 mmHg, a two-sided significance level of 5%, and a power of 80%. Based on these parameters, 34 participants are needed. Allowing for a 10% dropout rate, the final target sample size is set at 38 participants.

[Study Duration] From Institutional Review Board (IRB) approval to 18 months thereafter.

[Study Parameters]

* Demographics: age, sex, height, weight, body mass index, smoking status (current/ex/non), smoking pack-years
* Arterial blood gas analysis (3 times: baseline, crossover, end of study): pH, PaCO2, PaO2, HCO3-, SPO2
* PtCO2 (transcutaneous CO2)
* Pulmonary function test (within the last year): FEV1 (L), % predicted FEV1, FVC (L), % predicted FVC, FEV1/FVC (%)
* Dyspnea scale: mMRC score
* Home oxygen therapy status and flow rate
* Current treatment medications: inhaled bronchodilators, inhaled corticosteroids
* Average daily usage time

[Study Methods] Participants will be randomly assigned to NIV (Trilogy Evo®) or HFNC (myAirvo2®) in a 1:1 ratio for six weeks, then crossover to the alternate device for another six weeks. Assessments will be conducted at baseline (V1), after the first device (V2), and after crossover completion (V3).

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 40 years or older
* Diagnosed with COPD
* Arterial blood gas test, pCO2 > 45 mmHg at stable status
* A person who can read or write in Korean
* Written informed consent to participate in this study

Exclusion Criteria:

* A person who disagrees with the content of a informed consent
* Those who have difficulty wearing NIV or HFNC
* Cognitive impairment or apsychiatric disorder
* Hypoxic or hypercapnic exacerbation within the previous four weeks

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 38 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
PaCO2 | The first measurement will be conducted at baseline, on the day the first device is applied. The second measurement will be taken at week 6 from baseline, after the device has been used for six weeks. The final measurement will be performed at week 12 fr
  Arterial blood gas analysis will be performed three times to assess the improvement of hypercapnia, the primary outcome, by measuring pH, PaCO₂, PaO₂, HCO₃-, and SpO₂.

SECONDARY OUTCOMES:
TCO2 | The first measurement will be conducted at baseline, on the day the first device is applied. The second measurement will be taken at week 6 from baseline, after the device has been applied for six weeks. The final measurement will be performed at week 12
  Transcutaneous CO₂ (SenTec V-Sign, SenTec AG, Switzerland) will be measured three times as a surrogate marker for hypercapnia.
Compliance | The first assessment will be conducted at week 6 from baseline, after the first device has been applied for six weeks. The second assessment will be performed at week 12 from baseline, after the second device has been applied for six weeks.
  During the six-week application period of each device, the actual average daily usage time and the percentage of days with at least four hours of usage (number of days with ≥4 hours of use/ total number of applied days) ×100 will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Wonju Severance Christian Hospital, Wŏnju, Gangwondo, South Korea

IPD SHARING:
Plan to Share IPD: No